CLINICAL TRIAL: NCT04500652
Title: Evaluation of Mental Health Status and Related Factors Among Physical Medicine & Rehabilitation Physicians During the Covid-19 Pandemic
Brief Title: Mental Health Status and Related Factors Among Physical Medicine & Rehabilitation Physicians in the Covid-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Banu Dilek, Principal Investigator, Dokuz Eylul University
Other Study IDs: PMRMentalcovid
Record Dates: First submitted 2020-07-24; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Anxiety; Depression; Insomnia; Covid19; Coronavirus
Keywords: depression; anxiety; insomnia; Covid-19; coronavirus
MeSH Terms: conditions — Anxiety Disorders; Depression; Sleep Initiation and Maintenance Disorders; COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In December 2019, a highly infectious disease caused by a novel coronavirus (SARS-CoV-2) emerged in Wuhan, China. On March 11th 2020, the World Health Organization (WHO) declared COVID-19 a pandemic. Facing this critical situation, health care workers on the front line are at risk of developing psychological distress and other mental health symptoms. Physical medicine and rehabilitation (PM&R) physicians works both in specialty outpateint/inpatient clinic and pandemic outpatient/inpatient clinics during the outbreak. Accordingly, PM&R physicians are expected to be mentally affected by COVID-19 pandemic. In this study we aimed to evaluate mental health status of PM&R physicians and related factors during COVID-19 pandemic. This study is a cross-sectional survey which is conducted on an online platform. Demographic data, working conditions of PM&R physicians and factors that may be related to mental health status is questioned in the survey. The Depression, Anxiety and Stress Scale - 21 (DASS-21) is used to measure the emotional states of depression, anxiety and stress.The Insomnia Severity Index (ISI) is used to assess the severity of both nighttime and daytime components of insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Being a physical medicine and rehabilitation physician
* Worked during COVID-19 pandemic in specialty outpatient/inpatient clinic or pandemic outpatient/inpatient clinic.

Exclusion Criteria:

* Being a specialist in a branch other than physical medicine and rehabilitation

Ages: 24 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physical medicine and rehabilitation physicians in Turkey who worked during COVID-19 pandemic in specialty outpatient/inpatient clinic or pandemic outpatient/inpatient clinic.
Sampling Method: Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2020-06-27 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Depression, Anxiety and Stress Scales 21 Score | 5 months
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress.
Insomnia severity index score | 5 months
  The Insomnia Severity Index (ISI) is a brief instrument that was designed to assess the severity of both nighttime and daytime components of insomnia.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No